CLINICAL TRIAL: NCT03138148
Title: Evaluation of the Patient-ventilator Asynchrony During Mechanical Ventilation for Pediatric Acute Respiratory Failure
Acronym: Asynchrony
Status: Completed | Type: Observational
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Dr Guillaume Emeriaud, Principal Investigator, Intensivist, Clinical Associate Professor, St. Justine's Hospital
Other Study IDs: CHUSJ-3113
Record Dates: First submitted 2017-04-27; First posted 2017-05-03 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Mechanical Ventilation
Keywords: intensive care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Severe patient-ventilator asynchrony: Patients in whom the total percentage of time spent in asynchrony is superior to the entire cohort's 75th percentile
  Interventions: Other: Routine mechanical ventilation
- less severe patient-ventilator asynchrony: Patients in whom the total percentage of time spent in asynchrony is inferior to the entire cohort's 75th percentile
  Interventions: Other: Routine mechanical ventilation

INTERVENTIONS:
Other: Routine mechanical ventilation — Routine mechanical ventilation in PICU amid children with acute respiratory failure

SUMMARY:
The synchronization between the patient and the ventilator is an essential objective during mechanical ventilation (MV). Maintaining the patient's respiratory activity during MV reduces ventilation pressures, improves oxygenation, and decreases sedation. In order to do this, the inspiratory or expiratory effort of the patient must be detected by the respirator' sensor systems, so that the assistance delivered by the respirator is coordinated with the patient's respiratory cycles. The usual systems do not actually detect the beginning of the effort but its result: variation in flow rate or pressure at the respirator circuit, which depends on the patient's respiratory mechanics and sensitivity of the sensor. This detection is currently imperfect, which generates asynchrony between the patient's needs and the assistance of the respirator. The asynchrony comprises the periods of delay between the beginning of the inspiration (or expiration) and the response of the respirator, but also of the unsuitable cycles: inspiratory efforts of the patient not detected by the respirator, or inversely triggering assistance in the absence of inspiration by the patient (self-initiation), or delivery of 2 cycles of assistance for a single inspiration (double triggering).

Asynchrony is a risk factor for prolonged mechanical ventilation in adults. Adult studies have shown that patient-ventilator asynchrony is common during MV, and is associated with prolonged MV duration. An association with length of stay in intensive care and in hospital was also observed. In children, patient-ventilator synchronization is more difficult to achieve than in adults due to a higher respiratory rate and smaller current volumes. The impact of patient-ventilator asynchrony on evolution has not been studied in pediatrics.

Patient-ventilator synchronization could be improved by the development of new ventilatory modes. The new NAVA (neurally adjusted ventilatory assist) ventilation mode detects the patient's breathing efforts earlier by monitoring the electrical activity of the diaphragm through the esophagus. This new mode seems to improve synchronization in children. NAVA ventilation may therefore be a step forward, but its clinical benefits remain to be seen.

The objective of this study is to evaluate the impact of patient-ventilator asynchrony on the duration of mechanical ventilation in children with acute respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical ventilation planned for more than 24h according to the physician in charge;
* Presence of a spontaneous respiratory activity (defined by the presence of respiratory cycles activated by the patient);
* Parental consent obtained with the parents or with the legal representative.

Exclusion Criteria:

* pathologies for which a long and difficult weaning of the mechanical ventilation is expected: chronic respiratory failure with history of ventilation superior to one month, severe neurological or muscular pathology;
* Patients with a tracheotomy;
* Patients receiving a treatment by curare;
* Contraindication of recording of the diaphragmatic activity by oesophageal way, in particular recent oesophageal surgery, oesophageal stenosis, suspicion of diaphragmatic paralysis, severe coagulation disorder;
* Patients to whom a death seems imminent;
* Patients for whom a limitation of the care was considered.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients under mechanical ventilation for acute respiratory failure
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-05-26 (Actual); Primary Completion 2012-10-17 (Actual); Study Completion 2017-01-06 (Actual)

PRIMARY OUTCOMES:
Difference in ventilator free days | 28 days
  Difference in ventilator free days at Day 28th between the two patient groups (high versus moderate asynchrony)

SECONDARY OUTCOMES:
The impact of asynchrony on Comfort scale | at inclusion
  Comfort Scale between the two patient groups (high versus moderate asynchrony)
Intensive care unit length of stay | 28 days
  between the two patient groups (high versus moderate asynchrony)
Mortality in pediatric intensive care unit | 28 days
  between the two patient groups (high versus moderate asynchrony)

CONTACTS AND LOCATIONS:
Locations (1):
- St. Justine's Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No